CLINICAL TRIAL: NCT03554317
Title: COMbination of Bipolar Androgen Therapy and Nivolumab in Patients With Metastatic Castration-Resistant Prostate Cancer
Brief Title: COMbination of Bipolar Androgen Therapy and Nivolumab
Acronym: COMBAT-CRPC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J1812; IRB00164973 (Other: JHM IRB)
Record Dates: First submitted 2018-05-23; First posted 2018-06-13 (Actual); Results first posted 2023-10-03 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Castration-resistant Prostate Cancer; Metastatic Prostate Cancer; Prostate Cancer
Keywords: Bipolar Androgen Therapy; Testosterone; Nivolumab
MeSH Terms: conditions — Prostatic Neoplasms | interventions — testosterone 17 beta-cypionate; Testosterone Propionate; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Bipolar Androgen Therapy + Nivolumab (Experimental): All participants must have a rising PSA and/or radiographic progression and prior treatment with at least one novel androgen receptor (AR) targeted therapy (i.e. abiraterone acetate, enzalutamide). Up to one taxane agent for metastatic castration-resistant prostate cancer is permitted. Patients will be treated with testosterone cypionate 400mg IM every 4 weeks for a lead-in period of 12 weeks. After the lead-in period, all patients will be treated with nivolumab 480mg IV every 4 weeks and maintained on testosterone cypionate 400mg IM every 4 weeks. Treatment [with a minimum drug exposure of 12 weeks] will be continued until PSA progression (PCGW3 criteria) or clinical/radiographic progression (whichever comes first), or until unmanageable toxicity requiring drug cessation.
  Interventions: Drug: Testosterone cypionate; Drug: Nivolumab

INTERVENTIONS:
Drug: Testosterone cypionate — Depot (DEPO)-Testosterone Injection, for intramuscular (IM) injection, contains testosterone cypionate which is the oil-soluble 17 (beta)-cyclopentylpropionate ester of the androgenic hormone testosterone. Testosterone cypionate is a white or creamy white crystalline powder, odorless or nearly so and stable in air. Depot (DEPO)-Testosterone Injection is available in two strengths, 100 mg/mL and 200 mg/mL testosterone cypionate.
  Other Names: Depot (DEPO)-Testosterone Injection
Drug: Nivolumab — Nivolumab Injection, 100 mg/10 mL (10 mg/mL) or 40 mg/4 mL (10 mg/mL), is a clear to opalescent, colorless to pale yellow liquid, which may contain light (few) particulates. The drug product is a sterile, non-pyrogenic, single-use, isotonic aqueous solution formulated at 10 mg/mL in sodium citrate, sodium chloride, mannitol, diethylenetriaminepentacetic acid (pentetic acid), and polysorbate 80 (Tween 80), at potential hydrogen (pH) 6.0 and includes an overfill to account for vial, needle, and syringe holdup. It is supplied in 10-cc Type I flint glass vials, stoppered with butyl rubber. The clinical study product is a sterile solution to be administered through parenteral intravenous infusion.
  Other Names: BMS-936558; MDX1106; ONO-4538

SUMMARY:
Single arm, multicenter, open-label Phase II study of the effects of parenteral testosterone in combination with nivolumab in men with metastatic castration-resistant prostate cancer who previously progressed on at least one novel androgen-receptor targeted therapy (i.e. Abiraterone acetate, Enzalutamide). Up to one taxane agent is permitted.

DETAILED DESCRIPTION:
The trial will enroll up to 44 participants (45 were enrolled because the last two patients consented at two sites simultaneously). Eligible participants will continue on androgen ablative therapy with a GnRH analogue (i.e. Zoladex, Trelstar, Eligard, or Lupron) if they have not undergone orchiectomy. Following enrollment, participants will receive an intramuscular injection of testosterone cypionate 400mg every 4 weeks for a lead-in period of 12 weeks. After the lead-in period, all participants will be treated with nivolumab 480mg IV every 4 weeks and maintained on testosterone cypionate 400mg IM every 4 weeks. Assessments for response to testosterone + nivolumab will be performed approximately every 3 months. Treatment [with a minimum drug exposure of 12 weeks] will be continued until PSA progression (Prostate Cancer Working Group 3 [PCWG3] criteria) or clinical/radiographic progression (whichever comes first), or until unmanageable toxicity requiring drug cessation.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide signed informed consent.
* Males aged 18 years of age and above.
* Histological or cytologic proof of adenocarcinoma of the prostate.
* Known castration-resistant disease, defined according to Prostate Cancer Working Group 3 (PCWG3) criteria as:

  * Castrate serum testosterone level: ≤ 50 ng/dL (≤ 1.7 nmol/L).
  * Subjects who have failed initial hormonal therapy, either by orchiectomy or by using a gonadotropin-releasing hormone (GnRH) agonist in combination with an anti-androgen, must first progress through anti-androgen withdrawal prior to being eligible. The minimum time frame to document failure of anti-androgen withdrawal will be four weeks.
  * Serum Prostate Specific Antigen (PSA) progression defined as two consecutive increases in PSA over a previous reference value within 6 months of first study treatment, each measurement at least one week apart.

Or

* Documented bone lesions by the appearance of ≥ 2 new lesions by bone scintigraphy or dimensionally-measureable soft tissue metastatic lesion assessed by CT or MRI.

  * Absolute PSA ≥ 2.0 ng/mL at screening.
  * Must have PSA and/or radiographic progression on AT LEAST 1 novel AR targeted therapy (abiraterone acetate, enzalutamide). One prior chemotherapy agent for metastatic castration-resistant prostate cancer (mCRPC) will be allowed.
  * Prior treatment with abiraterone, enzalutamide, bicalutamide, and/or ketoconazole is allowed. There is no limit on the maximum number or types of prior hormonal therapies received.
  * Must be maintained on a GnRH analogue or have undergone orchiectomy.
  * Radiographic evidence of metastatic disease by CT scan and bone scan, performed within the prior 4 weeks.
  * Must have a soft tissue metastatic lesion available for biopsy collection to perform tumor tissue analysis.
  * Karnofsky Performance Status (KPS): ≥ 70% within 14 days before start of study treatment (ECOG ≤ 2).
  * Participants must have normal organ and bone marrow function measured within 28 days prior to administration of study treatment as defined below:
* Hemoglobin ≥ 9.0 g/dL with no blood transfusion in the past 28 days.
* Absolute neutrophil count (ANC) ≥ 1.0 x 10^9/L
* Platelet count ≥ 100 x 10^9/L
* Total bilirubin within institutional upper limit of normal (ULN) (In patients with Gilbert's syndrome, total bilirubin < 1.5x institutional ULN will be acceptable).
* Aspartate aminotransferase (AST) (Serum Glutamic Oxaloacetic Transaminase (SGOT)) / Alanine aminotransferase (ALT) (Serum Glutamic Pyruvate Transaminase (SGPT)) within institutional upper limit of normal.
* Participants must have creatinine clearance estimated ≥ 40 mL/min.

  * Participants must have a life expectancy ≥ 6 months.
  * Male participants and their partners, who are sexually active and of childbearing potential, must agree to the use of two highly effective forms of contraception in combination, throughout the period of taking study treatment and for 7 months after the last dose of nivolumab to prevent pregnancy in a partner.
  * No evidence (within 5 years) of prior malignancies (except successfully treated basal cell or squamous cell carcinoma of the skin).

Exclusion Criteria:

* Has received external-beam radiotherapy within the last 2 weeks prior to start of study treatment.
* Prior oral anti-androgen (e.g. bicalutamide, nilutamide, enzalutamide, apalutamide), or androgen synthesis inhibitor (e.g. abiraterone, orteronel) within the past 2 weeks is not permitted. 5-alpha reductase inhibitor therapy (e.g. finasteride, dutasteride) is allowed, as long as subject has been stable on medication for past 6 months.
* Prior treatment with chemotherapy for the treatment of metastatic hormone sensitive prostate cancer is allowed if the last dose of chemotherapy was greater than 6 months prior to enrollment. In addition, one chemotherapy agent for mCRPC will be allowed.
* Patients who have received prior treatment with bipolar androgen therapy (e.g. testosterone, BAT) are excluded.
* Pain due to metastatic prostate cancer requiring opioid therapy.
* Patients with an intact prostate AND urinary obstructive symptoms are excluded (which includes patients with urinary symptoms from benign prostatic hyperplasia (BPH)).
* Patients receiving anticoagulation therapy with Coumadin are not eligible for study. (Patients on non-coumadin anticoagulants (Lovenox, Xarelto, etc.) are eligible for study. Patients on Coumadin who can be transitioned to Lovenox or Xarelto prior to starting study treatments will be eligible).
* Patients with prior history of an arteriovenous thromboembolic event within the last 12 months are excluded.
* Patients allergic to sesame seed oil or cottonseed oil are excluded.
* Involvement in the planning and/or conduct of the study (applies to both BMS staff and/or staff at the study site).
* Participation in another clinical study with an investigational product during the last 4 weeks/28 days.
* Patients should be excluded if they have had prior systemic treatment with an anti-Programmed Cell Death Protein (PD)-1, anti-PD-L1, anti-PD-L2, anti-Cytotoxic T-lymphocyte-Associated Protein (CTLA)-4 antibody, or any other antibody or drug specifically targeting T-cell costimulation or immune checkpoint pathways (e.g. immune checkpoint antagonists).
* Evidence of disease in sites or extent that, in the opinion of the investigator, would put the patient at risk from therapy with testosterone (e.g. femoral metastases with concern over fracture risk, severe and extensive spinal metastases with concern over spinal cord compression, extensive liver metastases).
* Concurrent use of other anticancer agents or treatments, with the following exceptions:

  * Ongoing treatment with leutinizing hormone-releasing hormone (LHRH) agonists or antagonists, denosumab (Prolia) or bisphosphonate (e.g. zoledronic acid) is allowed. Ongoing treatment should be kept at a stable schedule; however, if medically required, a change of dose, compound, or both is allowed.
* Any treatment modalities involving major surgery within 4 weeks prior to the start of study treatment.
* Symptomatic nodal disease, i.e. scrotal, penile or leg edema (≥ CTCAE Grade 3).
* Patients are excluded if they have active known brain metastases or leptomeningeal metastases. Subjects with brain metastases are eligible if metastases have been treated and there is no magnetic resonance imaging (MRI) evidence of progression for at least 4 weeks after treatment is complete and within 28 days prior to the first dose of testosterone administration. There must also be no requirement for immunosuppressive doses of systemic corticosteroids (> 10 mg/day prednisone equivalents) for at least 2 weeks prior to study drug administration.
* Patients should be excluded if they have an active, known or suspected autoimmune disease (e.g. inflammatory bowel disease, rheumatoid arthritis, autoimmune hepatitis, lupus, celiac disease). Subjects are permitted to enroll if they have vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger.
* Patients should be excluded if they have a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration. Inhaled or topical steroids and adrenal replacement doses > 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease.
* Permitted therapies include topical, ocular, intra-articular, intranasal, and inhalational corticosteroids (with minimal systemic absorption). Physiologic replacement doses of systemic corticosteroids are permitted, even if > 10 mg/day prednisone equivalents. A brief course of corticosteroids for prophylaxis (e.g. contrast dye allergy) or for treatment of non-autoimmune conditions (e.g. delayed-type hypersensitivity reaction caused by contact allergen) is permitted.
* As there is potential for hepatic toxicity with nivolumab, drugs with a predisposition to hepatotoxicity should be used with caution in patients treated with nivolumab-containing regimen.
* Patients should be excluded if they have a positive test for hepatitis B virus surface antigen (HBV sAg) or hepatitis C virus ribonucleic acid (HCV antibody) indicating acute or chronic infection.
* Patients should be excluded if they have known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS).
* History of allergy to study drug components.
* History of severe hypersensitivity reaction to any monoclonal antibody.
* Other primary tumor (other than CRPC) including hematological malignancy present within the last 5 years (except non-melanoma skin cancer or low-grade superficial bladder cancer).
* Has imminent or established spinal cord compression based on clinical findings and/or MRI.
* Any other serious illness or medical condition that would, in the opinion of the investigator, make this protocol unreasonably hazardous, including, but not limited to:

  * Any uncontrolled major infection.
  * Cardiac failure New York Heart Association (NYHA) Class III or IV.
  * Crohn's disease or ulcerative colitis.
  * Bone marrow dysplasia.
  * Known allergy to any of the compounds under investigation.
  * Unmanageable fecal incontinence.
* Persistent toxicities (> CTCAE Grade 2) caused by previous cancer therapy, excluding alopecia.
* Poor medical risk due to a serious, uncontrolled medical disorder, non-malignant systemic disease or active, uncontrolled infection. Examples include, but are not limited to, uncontrolled ventricular arrhythmia, recent (within 6 months) myocardial infarction, uncontrolled major seizure disorder, extensive interstitial bilateral lung disease, or any psychiatric disorder that prohibits obtaining informed consent.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2018-09-05 (Actual); Primary Completion 2022-10-27 (Actual); Study Completion 2023-01-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Markowski, MD, Ph.D, Principal Investigator — Johns Hopkins University
Locations (3):
- United States (3):
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Markowski MC, Taplin ME, Aggarwal R, Sena LA, Wang H, Qi H, Lalji A, Sinibaldi V, Carducci MA, Paller CJ, Marshall CH, Eisenberger MA, Sanin DE, Yegnasubramanian S, Gomes-Alexandre C, Ozbek B, Jones T, De Marzo AM, Denmeade SR, Antonarakis ES. Bipolar androgen therapy plus nivolumab for patients with metastatic castration-resistant prostate cancer: the COMBAT phase II trial. Nat Commun. 2024 Jan 2;15(1):14. doi: 10.1038/s41467-023-44514-2. PMID 38167882

RESULTS

PARTICIPANT FLOW:
Groups:
- Bipolar Androgen Therapy + Nivolumab: All participants must have a rising PSA and/or radiographic progression and prior treatment with at least one novel androgen receptor (AR) targeted therapy (i.e. abiraterone acetate, enzalutamide). Up to one taxane agent for metastatic castration-resistant prostate cancer is permitted. Patients will be treated with testosterone cypionate 400mg IM every 4 weeks for a lead-in period of 12 weeks. After the lead-in period, all patients will be treated with nivolumab 480mg IV every 4 weeks and maintained on testosterone cypionate 400mg intramuscular (IM) every 4 weeks. Treatment [with a minimum drug exposure of 12 weeks] will be continued until PSA progression (PCGW3 criteria) or clinical/radiographic progression (whichever comes first), or until unmanageable toxicity requiring drug cessation.
Period: Overall Study
Arm/Group | Bipolar Androgen Therapy + Nivolumab
Started | 45
Completed | 37
Not Completed | 8
Not completed — Withdrawal by Subject | 1
Not completed — PSA Progression | 3
Not completed — Radiographic Progression | 4

BASELINE CHARACTERISTICS:
Arm/Group | Bipolar Androgen Therapy + Nivolumab
Number analyzed (Participants) | 45
Age, Continuous [Median (Full Range); unit: years] | 69 [51 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 45
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 40
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 45
Baseline PSA (ng/mL) [Median (Full Range); unit: ng/mL] — Prostate-specific antigen, or PSA, is a protein produced by normal, as well as malignant, cells of the prostate gland. The PSA test measures the level of PSA in the blood. For this test, a blood sample is sent to a laboratory for analysis. The results are usually reported as nanograms of PSA per milliliter (ng/mL) of blood.
  ng/mL | 57.6 [5.4 to 457]
Gleason sum [Count of Participants; unit: Participants] — For most prostate cancers, the Gleason sum ranges from 6 to 10. Gleason 6 is the least aggressive cancer type. Gleason 7 is intermediately aggressive. Gleason 8-10 is the most aggressive cancer type.
  Participants
    ≤ 7 | 11
    8 | 8
    9 | 18
    10 | 5
    Unknown | 3
Visceral disease [Count of Participants; unit: Participants] — Visceral disease is described as the presence of soft tissue lesions.
  Participants
    Yes | 7
    No | 38
Lines of Prior Novel AR (androgen receptor) Targeted Therapy [Count of Participants; unit: Participants]
  1 | 21
  ≥2 | 24
Prior Taxane Chemotherapy [Count of Participants; unit: Participants]
  Yes | 20
  No | 25
≥2 Novel AR (Androgen Receptor) Targeted Therapy and Prior Taxane Chemotherapy [Count of Participants; unit: Participants]
  Yes | 15
  No | 30

OUTCOME MEASURES:

1. Primary Outcome: Prostate Specific Antigen (PSA) Response to Bipolar Androgen Therapy + Nivolumab
Description: Number of participants with PSA response to Bipolar Androgen Therapy + Nivolumab. PSA response is counted for participants with ≥ 50% decline in PSA from baseline.
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Bipolar Androgen Therapy + Nivolumab
Number analyzed (Participants) | 45
Participants | 18

2. Secondary Outcome: Safety of Bipolar Androgen Therapy + Nivolumab As Determined by the Number of CTCAEs ≥ Grade 3
Description: Number of participants that experience adverse events grade ≥ 3, as defined by Common Terminology Criteria for Adverse Events (CTCAE).
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Bipolar Androgen Therapy + Nivolumab
Number analyzed (Participants) | 45
Participants | 5

3. Secondary Outcome: PSA Progression-Free Survival (PSA-PFS) to Bipolar Androgen Therapy + Nivolumab
Description: Number of months from the time of initiation on Bipolar Androgen Therapy + Nivolumab therapy until PSA increase of 25% over a nadir value, confirmed by a follow-up PSA at least 4 weeks apart.
Time Frame: 2 years
Measure: Number (95% Confidence Interval); unit: months
Arm/Group | Bipolar Androgen Therapy + Nivolumab
Number analyzed (Participants) | 45
months | 4.0 [3.6 to 5.0]

4. Secondary Outcome: Progression-Free Survival (PFS) to Bipolar Androgen Therapy + Nivolumab
Description: Median number of months from the time of the first dose to objective radiographic tumor progression or death, whichever comes first, as defined by RECIST 1.1 Criteria for progressive disease or death.
Time Frame: 2 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bipolar Androgen Therapy + Nivolumab
Number analyzed (Participants) | 45
months | 5.6 [5.4 to 6.8]

5. Secondary Outcome: Objective Response Rate (ORR) to Bipolar Androgen Therapy + Nivolumab
Description: Percentage of patients achieving a complete or partial response in target lesions as defined by RECIST 1.1 Criteria.
Time Frame: 2 years
Measure: Number; unit: percentage of overall participants
Arm/Group | Bipolar Androgen Therapy + Nivolumab
Number analyzed (Participants) | 45
percentage of overall participants | 18

6. Secondary Outcome: Durable Progression-Free Survival (Durable PFS) to Bipolar Androgen Therapy + Nivolumab
Description: Number of participants without clinical/radiographic progression for > 6 months from the start of treatment.
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Bipolar Androgen Therapy + Nivolumab
Number analyzed (Participants) | 45
Participants | 15

7. Secondary Outcome: Median Overall Survival (OS) to Bipolar Androgen Therapy + Nivolumab
Description: Median number of months from study enrollment to death from any cause up to 2 years after the last dose of study treatment received.
Time Frame: 3 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bipolar Androgen Therapy + Nivolumab
Number analyzed (Participants) | 45
months | 24.4 [17.6 to 31.1]

8. Other Pre Specified Outcome: PSA Response to Bipolar Androgen Therapy + Nivolumab in Patients With Gene Mutations
Description: Number of patients with ≥ 50% decline in PSA from baseline in patients with a somatic or germline mutation in homologous repair (HR) and/or mismatch repair (MMR) genes.
Time Frame: 2 years
Reporting Status: Not Posted

9. Other Pre Specified Outcome: PSA Response to Bipolar Androgen Therapy + Nivolumab in Patients Without Gene Mutations
Description: Number of patients with ≥ 50% decline in PSA from baseline in patients without a somatic or germline mutation in homologous repair (HR) and/or mismatch repair (MMR) genes.
Time Frame: 2 years
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Clinical Response Association of Bipolar Androgen Therapy + Nivolumab to Mutation-associated Neoantigens (MANAs).
Description: Clinical Response Association of Bipolar Androgen Therapy + Nivolumab to mutation-associated neoantigens (MANAs) can be assessed by the number of patients treated with Bipolar Androgen Therapy + Nivolumab with the presence of MANAs.
Time Frame: 3 years
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Clinical Response Association to Bipolar Androgen Therapy + Nivolumab as Assessed by the Generation of Tumor-associated Neoantigens (TAAs)
Description: Clinical Response Association to Bipolar Androgen Therapy + Nivolumab with generation of tumor-associated neoantigens (TAAs) can be assessed by the number of patients treated with Bipolar Androgen Therapy + Nivolumab that have TAAs.
Time Frame: 3 years
Reporting Status: Not Posted

12. Other Pre Specified Outcome: PSA Correlation With Immune Markers in Response to Bipolar Androgen Therapy + Nivolumab
Description: Immunohistochemistry (IHC) staining will be used to quantify the number of immune markers present in pre-treatment and on-treatment biopsies in responders whose PSA has declined ≥ 50% versus non-responders.
Time Frame: 2 years.
Reporting Status: Not Posted

13. Other Pre Specified Outcome: PSA Correlation With DNA Damage Markers in Response to Bipolar Androgen Therapy + Nivolumab
Description: Immunohistochemistry (IHC) staining will be used to quantify the number of DNA damage markers present in pre-treatment and on-treatment biopsies in responders whose PSA has declined ≥ 50% versus non-responders.
Time Frame: 2 years.
Reporting Status: Not Posted

14. Other Pre Specified Outcome: Correlation of Bipolar Androgen Therapy on the Production of Inflammatory Chemokines and Cytokines
Description: Milliplex human cytokine/chemokine Immunology Multiplex Assay (Millipore-Sigma) will be used to assay acute effects of Bipolar Androgen Therapy by detecting the amount of cytokines and chemokines produced during therapy.
Time Frame: 2 years.
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse events were assessed up to 2 years. All-Cause Mortality was assessed up to 3 years
Arm/Group | Bipolar Androgen Therapy + Nivolumab
All-Cause Mortality (participants affected / at risk) | 13/45
Serious Adverse Events (participants affected / at risk) | 11/45
Other Adverse Events (participants affected / at risk) | 45/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bipolar Androgen Therapy + Nivolumab (N=45)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Chest pain - cardiac (Cardiac disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Fever (General disorders) | 2 (2)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Investigations - Other, abnormal ECG (Investigations) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 1 (2)
Lung infection (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2)
Pain in extremity (General disorders) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1)
Pericarditis (Cardiac disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1)
Rectal fistula (Gastrointestinal disorders) | 1 (1)
Renal and urinary disorders - Other, left-sided renal obstruction (Renal and urinary disorders) | 1 (1)
Urinary tract infection (Renal and urinary disorders) | 2 (2)
Vascular disorders - Other, deep vein thrombosis (Vascular disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Blood lactate dehydrogenase increased (Blood and lymphatic system disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bipolar Androgen Therapy + Nivolumab (N=45)
Bloating (Gastrointestinal disorders) | 1 (45)
Abdominal pain (Gastrointestinal disorders) | 6 (6)
Respiratory, thoracic and mediastinal disorders - Other, acute hypoxic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Alanine aminotransferase increased (Investigations) | 4 (4)
Alkaline phosphatase increased (Investigations) | 2 (2)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Serum amylase increased (Investigations) | 1 (3)
Anemia (Blood and lymphatic system disorders) | 1 (4)
Edema limbs (General disorders) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (8)
Aspartate aminotransferase increased (Investigations) | 5 (5)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 14 (24)
Blood bilirubin increased (Investigations) | 2 (2)
Blurry vision (Eye disorders) | 1 (1)
Chest pain - cardiac (Cardiac disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 2 (3)
Constipation (Gastrointestinal disorders) | 10 (10)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (6)
CPK increased (Investigations) | 4 (5)
Creatinine increased (Investigations) | 7 (8)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 9 (11)
Dizziness (Psychiatric disorders) | 3 (3)
Dry mouth (Gastrointestinal disorders) | 1 (1)
Vascular disorders - Other, deep vein thrombosis (Vascular disorders) | 1 (1)
Dysgeusia (Nervous system disorders) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Dyspnea (Renal and urinary disorders) | 6 (6)
Edema face (General disorders) | 2 (2)
Edema limbs (General disorders) | 11 (15)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Conjunctivitis (Eye disorders) | 1 (1)
Eye disorders - other, double vision (Eye disorders) | 1 (1)
Flushing (Vascular disorders) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 2 (2)
Fatigue (General disorders) | 10 (13)
Fever (General disorders) | 2 (3)
Flu like symptoms (General disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (2)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Genital edema (Reproductive system and breast disorders) | 2 (2)
Hypertrichosis (Skin and subcutaneous tissue disorders) | 1 (1)
Headache (Nervous system disorders) | 3 (3)
Hematuria (Renal and urinary disorders) | 4 (4)
Hot flashes (Vascular disorders) | 1 (1)
Renal and urinary disorders - Other, hydrocalycosis (Renal and urinary disorders) | 1 (1)
Hyperglycemai (Metabolism and nutrition disorders) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1)
Hypertension (Vascular disorders) | 3 (4)
Hyperthyroidism (Endocrine disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (2)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (2)
Hypotension (Vascular disorders) | 1 (1)
Hypothyroidism (Endocrine disorders) | 5 (5)
Ileus (Gastrointestinal disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Investigations - Other, elevated white blood cells (Investigations) | 1 (1)
Irritability (Psychiatric disorders) | 5 (5)
Kidney infection (Renal and urinary disorders) | 1 (1)
Lipase increased (Investigations) | 4 (8)
Localized edema (General disorders) | 2 (2)
Lung infection (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Skin and subcutaneous tissue disorders - Other, macular rash (Skin and subcutaneous tissue disorders) | 1 (1)
Musculoskeletal and connective tissue disorders - other, restless legs (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 4 (5)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 4 (5)
Nausea (Gastrointestinal disorders) | 18 (19)
Non-cardiac chest pain (General disorders) | 2 (2)
Pain (General disorders) | 6 (13)
Pain in extremity (General disorders) | 14 (23)
Pneumontiis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (3)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (3)
Rectal fistula (Gastrointestinal disorders) | 1 (1)
Rectal pain (Gastrointestinal disorders) | 1 (1)
Renal and urinary disorders - Other, urinary dysfunction (Renal and urinary disorders) | 1 (1)
Serum amylase increased (Investigations) | 3 (4)
Sinusitis (Infections and infestations) | 1 (1)
Skin and subcutaneous tissue disorders - Other, macular rash (Skin and subcutaneous tissue disorders) | 3 (3)
Skin and subcutaneous tissue disorders - Other, pruritic rash (Skin and subcutaneous tissue disorders) | 1 (1)
Skin and subcutaneous tissue disorders - Other, follicular rash (Skin and subcutaneous tissue disorders) | 1 (1)
Skin infection (Skin and subcutaneous tissue disorders) | 1 (1)
Skin and subcutaneous tissue disorders - Other, desquamation (Skin and subcutaneous tissue disorders) | 1 (1)
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Spinal cord compression (Nervous system disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Testicular disorder (Reproductive system and breast disorders) | 1 (1)
Thrush (Infections and infestations) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 1 (1)
Tooth infection (Infections and infestations) | 1 (1)
Tremor (Nervous system disorders) | 1 (1)
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 3 (3)
Urinary incontinence (Renal and urinary disorders) | 3 (4)
Urinary retention (Renal and urinary disorders) | 3 (3)
Urinary tract infection (Renal and urinary disorders) | 1 (5)
Urinary tract obstruction (Renal and urinary disorders) | 1 (1)
Urinary urgency (Renal and urinary disorders) | 1 (1)
Uveitis (Eye disorders) | 1 (2)
Vertigo (Ear and labyrinth disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 7 (9)
Bone pain (Musculoskeletal and connective tissue disorders) | 3 (4)
Breast pain (Reproductive system and breast disorders) | 3 (3)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Facial pain (General disorders) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1)
Injection site reaction (General disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1)
Paresthesia (Nervous system disorders) | 1 (1)
Platelet count decreased (Investigations) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI may not publish results before Sponsor/Sponsor PI. If no multicenter publication within 12 months from study completion or termination at all sites, PI may publish results as long as Sponsor PI has copy of communication for review and comment at least 30 days before submission. Sponsor may request PI hold communication for additional 65 days to allow for filing of patent application or other methods to preserve proprietary and/or patent rights.

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-06-09): https://cdn.clinicaltrials.gov/large-docs/17/NCT03554317/Prot_SAP_000.pdf
  • Informed Consent Form (2020-10-06): https://cdn.clinicaltrials.gov/large-docs/17/NCT03554317/ICF_001.pdf